CLINICAL TRIAL: NCT02563184
Title: Seasonal Influenza Vaccine, Quadrivalent Versus Trivalent in Patients With Advanced Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Banner Health (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, David Baratz, M.D., Medical Doctor, Banner Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Flu Vaccine Quad vs Tri
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD (Active Comparator): Group will receive either the Fluzone Trivalent or Fluzone Quadrivalent.
  Interventions: Biological: Fluzone
- Control (Active Comparator): Group will receive either the Fluzone Trivalent or Fluzone Quadrivalent.
  Interventions: Biological: Fluzone

INTERVENTIONS:
Biological: Fluzone

SUMMARY:
To evaluate the magnitude of the humoral immune responses to quadrivalent vs trivalent influenza vaccines in adults between the age of 50 and 64 years with a prior diagnosis of GOLD Stage C and D COPD vs. those patients without COPD.

DETAILED DESCRIPTION:
Primary Objectives:

To evaluate the magnitude of the humoral immune responses to quadrivalent vs trivalent influenza vaccines in adults between the age of 50 and 64 years with a prior diagnosis of GOLD Stage C and D COPD (vs. those patients without COPD).

To demonstrate immunogenicity by measuring hemagglutination inhibiting antibodies (HI) against the components of viral antigens using seroconversion (≥4 fold increase over baseline titers) and sero-protection (HI titer of ≥40 against the vaccine components).

Secondary Objective:

To assess the degree of antibody response of COPD patients based on severity of disease as measured by FEV1.

To assess the impact of inhaled corticosteroids on the adaptive immune response after vaccination.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients with COPD will be:

1. Signed informed consent prior to initiation of study-mandated vaccination.
2. Patients with spirometric data in the preceding 18 months confirming the diagnosis of COPD.
3. Patients meeting GOLD Classification of Stage C or Stage D COPD.
4. Patients 50 years old - 64 years old.

Inclusion criteria for Healthy participants will be:

1. Signed informed consent prior to initiation of study-mandated vaccination.
2. No active symptoms of lung disease.
3. FEV1/FVC in the normal range > 70% age predicted value.
4. No history of tobacco use/abuse.
5. No prior history of alpha-1 antitrypsin deficiency.
6. Patients 50 years old - 64 years old.

Exclusion Criteria:

1. Severe allergy to eggs.
2. Severe reaction to past doses of influenza vaccine.
3. Guillian-Barre syndrome.
4. Currently recieving dialysis.
5. Current, active, treatment for cancer.
6. History of transplant (allograft).
7. Dementia or Alzheimer's disease diagnosis.
8. Prior diagnosis of HIV or AIDS.
9. Moderate to severe pulmonary hypertension.
10. Serum AST/ALT > 3x the upper limit of normal.
11. Patients with exacerbations or respiratory infection during the 4 weeks preceding the onset of the study.
12. Active pregnancy.
13. Systemic immunomodulating medications.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Hemagglutination inhibiting antibodies (HI) against the components of viral antigens | 3 months
  The investigators will be measuring hemagglutination inhibiting antibodies (HI) against the components of viral antigens using seroconversion (≥4 fold increase over baseline titers) and sero-protection (HI titer of ≥40 against the vaccine components)

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Associates, Phoenix, Arizona, United States